CLINICAL TRIAL: NCT07064733
Title: A Randomized Controlled Trial on the Effect of Music Therapy and Warm Foot Bath Therapy on Anxiety, Blood Pressure, and Quality of Life in Low-Risk Primigravida Pregnant Women
Brief Title: Effect of Music and Warm Foot Bath Therapy on Pregnancy-Related Anxiety, Blood Pressure and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Nermin Kayar, lecturer, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Trakya University
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Primigravida Women; Music Therapy; Blood Pressure Monitoring; Quality of Life; Anxiety
Keywords: primigravida; music therapy; Warm Foot Bath; Quality of Life; blood pressure
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four parallel groups: (1) music therapy only, (2) warm foot bath therapy only, (3) combined music and foot bath therapy, or (4) control group with no intervention. Each intervention group will receive their respective therapy for 2 weeks, 3 times per week. Pre- and post-intervention assessments of anxiety, blood pressure, and quality of life will be conducted. The control group will receive usual antenatal care without any intervention but will be assessed using the same outcome measures.
Masking Description: This study is open-label. Due to the nature of the interventions-music therapy and warm foot bath-it is not possible to blind participants or investigators. All participants and study staff are aware of the assigned intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- music therapy group (Experimental): At 26 weeks and above, low-risk primigravida pregnant women will be informed about the purpose of the study and voluntary participation will be ensured. Those who score 20 and above on both subscales of the State-Trait Anxiety Inventory will be included in the study. Participants will be educated about music therapy and blood pressure measurement at the first home visit and brochures will be provided. Contact information will be obtained and the EQ-5D General Quality of Life Scale will be applied. Handpan music rhythm with a volume level not exceeding 60 dB will be played for 30 minutes in the morning and evening, 3 days a week when the pregnant woman is available. Blood pressure measurements will be made before and after the session (0, 30, 60 minutes), and the scales will be reapplied by telephone at the end of the week. In pregnant women hospitalized in the ward, the same protocol will be applied by the coordinator during hospitalization.
  Interventions: Other: Music Therapy
- Warm water foot bath therapy group (Experimental): At 26 weeks and above, low-risk primigravida pregnant women hospitalized in outpatient clinic or obstetrics and gynecology service will be explained the purpose of the study and voluntary participation will be ensured. Those who score 20 and above on both subscales of the State-Trait Anxiety Inventory will be included in the study. During the first home visit, warm water foot bath (37-40°C, 10-15 min), education about the application and blood pressure measurement will be given and a brochure will be presented. Contact information will be obtained and the EQ-5D Quality of Life Scale will be applied. Foot baths will be applied 3 days a week, morning and evening, when the pregnant woman is available. Blood pressure measurements will be made before and after the session (0, 30, 60 minutes). At the end of the weeks, the scales will be repeated by telephone. For pregnant women hospitalized in the ward, the same protocol will be applied during hospitalization.
  Interventions: Other: warm water foot bath therapy
- Music therapy and foot bath group (Combine Group) (Experimental): At 26 weeks and above, low-risk primigravida pregnant women will be informed about the purpose of the study and voluntary participation will be ensured. Those who score 20 and above on both subscales of the State-Trait Anxiety Inventory will be included. During the first home visit, a brochure will be given about music therapy and warm water foot bath (37-40°C, 10-15 minutes). In music therapy, a quiet, dimly lit environment, appropriate position and positive thoughts will be suggested. Contact information of the pregnant woman will be obtained and EQ-5D Quality of Life Scale will be applied. A warm water foot bath will be taken in the morning and evening, 3 days a week, and then a handpan music recording will be played for 30 minutes at 60 dB. Blood pressure measurements will be made before and after the session (0, 30, 60 minutes). At the end of the weeks, the scales will be repeated by telephone. Pregnant women hospitalized in the ward will follow the same protocol.
  Interventions: Other: Music Therapy; Other: warm water foot bath therapy
- Control Group (No Intervention): At 26 weeks and above, low-risk primigravida pregnant women with outpatient follow-up or hospitalization in the obstetrics and gynecology service will be explained the purpose of the study and voluntary participation will be ensured. Pregnant women who scored 20 and above on both subscales of the State-Trait Anxiety Inventory will be included in the study. Blood pressure measurements will be made in the morning and evening on 3 days of the week, and the scales will be reapplied at the end of the first and second week. No intervention will be made to the pregnant women. At the end of the study, pregnant women in the control group will be offered optional music therapy and warm water foot baths.

INTERVENTIONS:
Other: Music Therapy — The music therapy intervention consists of listening sessions using specially recorded handpan music, designed to promote relaxation and reduce anxiety in pregnant women. The handpan is a melodic percussion instrument known for its soothing and harmonic sound qualities.
  Participants will listen to a 30-minute handpan music recording at home, in a quiet and dimly lit room, while resting in a semi-fowler or left lateral position. The sound volume will be kept below 60 decibels to ensure comfort and prevent overstimulation. Sessions will be scheduled three times per week, in the morning and evening, over a two-week period.
  Before each session, participants will be reminded by phone and instructed to measure their blood pressure immediately prior to and at 0, 30, and 60 minutes after the music listening. The therapy aims to create a calming environment that encourages positive thoughts and bonding with the fetus.
  Arms: Music therapy and foot bath group (Combine Group); music therapy group
Other: warm water foot bath therapy — The warm water foot bath therapy involves soaking the participant's feet in water heated to 37-40°C for 10-15 minutes per session. This therapy is designed to promote relaxation, improve peripheral circulation, and reduce anxiety symptoms.
  Participants will perform the foot bath in a safe and comfortable setting, ensuring water temperature is monitored with a thermometer before each session. After soaking, feet should be thoroughly dried to prevent slipping, and participants are advised to have a companion nearby when standing up to avoid falls.
  The intervention will be applied three times weekly, in the morning and evening, over a two-week period. Blood pressure measurements will be taken immediately before and at 0, 30, and 60 minutes after each session.
  Arms: Music therapy and foot bath group (Combine Group); Warm water foot bath therapy group

SUMMARY:
Study Title:

The Effects of Music Therapy and Warm Foot Bath on Pregnancy-Related Stress, Blood Pressure, and Quality of Life in Low-Risk Primigravida Women

Brief Summary:

This randomized controlled trial investigates the impact of music therapy and warm foot bath therapy on pregnancy-related anxiety, blood pressure levels, and quality of life in low-risk primigravida pregnant women. Participants will be randomly assigned into four groups: music therapy, warm foot bath therapy, combined therapy, and control group. The interventions will be carried out for 2 weeks with pre- and post-assessments of anxiety and quality of life.

DETAILED DESCRIPTION:
Pregnancy is a period of significant physiological and psychological changes that can increase anxiety levels in women. This study aims to assess whether non-pharmacological interventions such as music therapy (handpan music) and warm foot baths can reduce anxiety, regulate blood pressure, and improve the quality of life in low-risk primigravida pregnant women at 26 weeks of gestation and above. A total of 144 participants will be randomly assigned to one of four groups and followed for two weeks. Data collection tools will include the State-Trait Anxiety Inventory (STAI TX-1 and TX-2), blood pressure monitoring forms, and EQ-5D quality of life scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years of age,

  * Literate; able to make an informed decision to participate, communicate verbally, and sign a consent form
  * Pregnant with a single, live fetus
  * Have a smartphone
  * Low-risk primigravida pregnant with a gestational age of 26 weeks or more

Exclusion Criteria:

* - Having hearing impairment,
* Refusing to participate,
* Being illiterate,
* Having communication problems,
* Being hospitalized with severe preeclampsia,
* The newborn not surviving.
* Antepartum hemorrhage
* Preeclampsia,
* Gestational hypertension,
* Cervical insufficiency,
* Having pregnancy-related complications such as congenital fetal anomalies and intrauterine growth restriction diagnosed before 28 weeks of gestation or having multiple pregnancies;
* Having psychiatric disorders (known anxiety or depression, other illnesses),
* Having medical problems such as endocrine disorders (gestational diabetes mellitus, thyroid dysfunction, etc.);
* Having assisted reproductive techniques (ART) such as in vitro fertilization, embryo transfer, or
* Pregnant women at risk of preterm birth will not be included in the study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 144 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in State Anxiety Score | Baseline, Day 7, and Day 14
  It consists of two subscales of 20 items each measuring state and trait anxiety. The State Anxiety Inventory (SAI) asks the individual to describe how he/she feels at a particular moment and under certain conditions; the Trait Anxiety Inventory (TAI) asks the individual to describe how he/she feels in general. The inventory is rated on a 4-point scale. Higher scores indicate higher levels of anxiety. In Spielberger's State and Trait Anxiety Inventory, 0-19 points are considered as No Anxiety, 20-39 points as Mild Anxiety, 40-59 points as Moderate Anxiety, 60-79 points as Severe Anxiety and 80 points as Panic.
EQ-5D General Quality of Life Scale | Baseline, Day 7, and Day 14
  The scale is a short, generic instrument used to define quality of life and to assign a quantitative value to health status. It consists of a VAS scale (excellent health to death) and 5 3-choice questions (mobility, self-care, usual daily tasks, pain discomfort, anxiety demoralization). The answers to each item have 3 options: no problem, some problem and major problem. As a result, the scale identifies 243 possible different health outcomes. An index score ranging from -0.59 to 1 is calculated from the 5 dimensions of the scale. In the score function, a value of 0 indicates death, a value of 1 indicates perfect health, while negative values indicate conditions such as unconsciousness, living bedridden, etc.
blood pressure Measurement | Days 1, 3, 5, 8, 10, and 12; with measurements at pre-, immediate post-, 30-min post-, and 60-min post-intervention, morning and evening sessions.
  Systolic and diastolic blood pressure will be measured at rest using a standardized sphygmomanometer immediately before the intervention, and at 0, 30, and 60 minutes after the intervention sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified participant data, study protocols, and analysis plans will be made available upon reasonable request to qualified researchers following publication of the study results. Data sharing will comply with ethical guidelines and participant confidentiality will be strictly maintained.

REFERENCES:
- [Background] Soylu N, Bulbul T, Muderris II. The effect of music on fetal well-being and anxiety levels and vital signs of pregnant women during non-stress test: Turkey sample. Health Care Women Int. 2022 May;43(5):499-517. doi: 10.1080/07399332.2021.1973010. Epub 2021 Sep 14. PMID 34520324
- [Background] E Aksoy Y, D Yilmaz S, Kilic S. The effect of music therapy on non-stress test results and anxiety levels in high-risk pregnant women: A randomized controlled trial. Int J Nurs Pract. 2024 Dec;30(6):e13281. doi: 10.1111/ijn.13281. Epub 2024 Jun 20. PMID 39031663
- [Background] Estrella-Juarez F, Requena-Mullor M, Garcia-Gonzalez J, Lopez-Villen A, Alarcon-Rodriguez R. Effect of Virtual Reality and Music Therapy on the Physiologic Parameters of Pregnant Women and Fetuses and on Anxiety Levels: A Randomized Controlled Trial. J Midwifery Womens Health. 2023 Jan;68(1):35-43. doi: 10.1111/jmwh.13413. Epub 2022 Nov 16. PMID 36383473